CLINICAL TRIAL: NCT03303040
Title: The Effect of Intermittent Hemidiaphragm Stimulation During Surgery on Mitochondrial Function, Single Fiber Contractile Force and Catabolic Pathways in Humans
Brief Title: Effect of Diaphragm Stimulation During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Arizona (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB201602186-N; R01AR072328 (NIH)
Record Dates: First submitted 2017-09-26; First posted 2017-10-05 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Mechanical Ventilation Complication; Diaphragm Injury
Keywords: Mechanical ventilation; Diaphragm weakness; Difficulty weaning from mechanical ventilation; Diaphragm stimulation

STUDY DESIGN:
Intervention Model Description: This is a within subjects design. One side of each subject's diaphragm will be stimulated. The other side of the subject's diaphragm will not be stimulated and will therefore serve as the control. Biopsies will be taken from both sides and compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation (Experimental): Electrical stimulation of hemidiaphragm
  Interventions: Other: Electrical stimulation of hemidiaphragm
- Control (No Intervention): No stimulation of hemidiaphragm

INTERVENTIONS:
Other: Electrical stimulation of hemidiaphragm — Electrical impulses
  Arms: Stimulation

SUMMARY:
During major surgical procedures general anesthesia is used to make the patient unconscious. General anesthesia insures that the patient is unaware of any pain caused by surgery. General anesthesia also prevents the patient from moving to prevent any potential surgical error. At the same time general anesthesia makes it impossible for the patient to breathe. To help the patient breathe a breathing tube is placed into the patient's airway and connected to the mechanical ventilator. A mechanical ventilator is an artificial breathing pump, which delivers gas into a patient's airways.

The purpose of this research study is to determine if brief periods of diaphragm stimulation can prevent diaphragm problems caused by the use of mechanical ventilators and surgery. To answer this question the changes in the genes responsible for maintaining diaphragm function will be studied. A gene is the code present in each cell in your body and controls the behavior of that cell. In addition, the changes in the contractile properties of muscle fibers will be studied. The results from this study may help develop new treatments to prevent diaphragm weakness resulting from mechanical ventilation use.

DETAILED DESCRIPTION:
Although mechanical ventilation (MV) is life-sustaining, it comes with a cost. MV dramatically reduces diaphragm contractility, induces ventilator-induced diaphragm dysfunction (VIDD) and sometimes leads to weaning failure. VIDD includes reduced mitochondrial respiration and increased oxidative stress, muscle fiber damage and decreased diaphragm force production.

In animal models, intermittent diaphragm contraction during MV support attenuates VIDD. However, there are only limited data addressing this problem in humans. Here, the study team propose to directly test the hypothesis that intermittent electrical stimulation (ES) of the human hemidiaphragm during prolonged cardiac surgeries with MV support prevents/attenuates VIDD in the active hemidiaphragm. Mitochondrial function is central to energy metabolism and skeletal muscle function in a chronically active muscle, such as the diaphragm. Although abnormal mitochondrial function is thought to precipitate VIDD in animal models, limited data are available concerning mitochondrial contributions to VIDD in humans. Of even greater importance, there are no interventions available to attenuate these defects in humans. Here, the study team will test the impact of an innovative experimental treatment, intermittent electrical stimulation (ES) of the hemidiaphragm during prolonged surgeries with MV, on mitochondrial function, single fiber contractile properties and catabolic muscle pathways in human diaphragm. Using a within-subjects experimental design, muscle samples from a stimulated hemidiaphragms will be compared with samples from the unstimulated hemidiaphragm. The study team will investigate mitochondrial dysfunction and oxidative stress during prolonged CTS/MV, and the potential of ES to attenuate or prevent VIDD. Next, the study team will investigate the effects of ES on single fiber contractile properties and Titin integrity. Finally, the study team will study the effect of ES on proteolytic pathways (caspase, calpain and ubiquitin-proteasome) and ribosomal RNA markers of decreased protein synthesis implicated in VIDD.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing complex, elective prolonged surgeries, usually lasting 5-8 hours or longer, including lung transplants (e.g. valveoplasty, coronary artery bypass and/or aortic repairs)

Exclusion Criteria:

* history of prior surgery to the diaphragm or pleura;
* a diagnosis of COPD will be determined from a clinical history consistent with chronic bronchitis and/or emphysema, a long history of cigarette smoking, and pulmonary function tests consistent with irreversible airflow obstruction (FEV1 < 40% predicted, according to European Respiratory Society criteria [will not apply to transplant patients]
* a diagnosis of chronic heart failure (NYHA class IV)
* clinical diagnosis of other lung disease (cystic fibrosis, bronchiectasis, lung cancer; etc.) [will not apply to transplant patients]
* renal insufficiency (serum creatinine > 1.6 mg/dl);
* severe hepatic disease (any liver function tests > 1.5 times the upper limit of normal);
* undernourishment (body mass index < 20 kg/m2),
* chronic uncontrolled or poorly controlled metabolic diseases (e.g., diabetes, hypo- or hyperthyroidism)
* orthopedic diseases, suspected paraneoplastic or myopathic syndromes,
* if in the surgeons' judgment the patients' clinical status warrants, diaphragm stimulation will be stopped and biopsies will not be obtained,

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 12 females and 12 males (based on gender identity) will be recruited for the study
Enrollment: 25 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anatole D Martin, PhD, Principal Investigator — University of Florida; Thomas M Beaver, MD, Principal Investigator — University of Florida; Barbara Smith, PhD, PT, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Undergoing Elective, Open Cardiothoracic Surgical Procedures Lasting 4 Hours or Greater: Patients undergoing complex, elective prolonged surgeries, usually lasting 5-8 hours or longer, including lung transplants (e.g. valvuloplasty, coronary artery bypass and/or aortic repairs)
Period: Overall Study
Arm/Group | Participants Undergoing Elective, Open Cardiothoracic Surgical Procedures Lasting 4 Hours or Greater
Started | 25
Completed | 21
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Participants Undergoing Elective, Open Cardiothoracic Surgical Procedures Lasting 4 Hours or Greater
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: Number] | 59 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Number of stimulations [Mean (Standard Deviation); unit: Number of Stimulations] | 6.2 (1.9)
Stimulation Current Intensity [Mean (Standard Deviation); unit: mA] | 18.0 (5.4)
%Force Vital Capacity [Mean (Standard Deviation); unit: Percentage of predicted value] | 86.6 (14.4)
% Forced Expiratory Volume [Mean (Standard Deviation); unit: Percentage of predicted] | 83.2 (15.0)
Maximal Inspiratory Pressure [Mean (Standard Deviation); unit: cm H2O] — Maximal voluntary static contractions of the inspiratory muscles against a closed valve, measured at the mouth.
  cm H2O | 90.6 (23.0)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 29.8 (3.96)
Intubation to Biopsy [Mean (Standard Deviation); unit: Minutes] — Measurement of the amount of time in minutes between intubation and muscle biopsy acquisition
  Minutes | 278 (65)
Intubation to Frist Stimulation [Mean (Standard Deviation); unit: Minute] | 98 (33)
Cardiopulmonary Bypass [Mean (Standard Deviation); unit: Minutes] | 137 (65)
Minimum Core Temperature [Mean (Standard Deviation); unit: Degrees Celsius] | 33.5 (2.4)
Core Temperature at Biopsy [Mean (Standard Deviation); unit: Degrees Celsius] | 36.5 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Mitochondrial Respiration
Description: High-resolution respirometry will be used to assess mitochondrial respiration of permeablilized diaphragm bundles. Addition of substrate medium to the Oroboros O2K respirometry instrument enables quantification of leak respiration and peak uncoupled respiration, expressed as pmol oxygen/sec/mg wet weight.
Time Frame: Up to eight hours
Population: Mitochondrial respiration was measured in the stimulated (n=19) and unstimulated (n=19) hemidiaphragms from subjects who completed the entire intra-operative stimulation protocol. Biopsy tissue was specifically reserved for analysis. From the full patient sample, insufficient contractile tissue was available to measure mitochondrial respiration in two unstimulated and two stimulated hemidiaphragms.
Measure: Mean (Standard Deviation); unit: pmol/s/mg wwt
Arm/Group | Control | Stimulation
Number analyzed (Participants) | 19 | 19
pmol/s/mg wwt
  Leak Respiration | 3.5 (0.7) | 2.9 (0.6)
  ECI+II | 31.1 (3.5) | 27.1 (2.1)

2. Primary Outcome: Aconitase Activity
Description: In order to evaluate mitochondrial damage, actonitase activity will be measured spectrophotometrically. It will be quantified as units/mg protein.
Time Frame: Up to eight hours
Population: Aconitase activity was measured in the stimulated (n=20) and unstimulated (n=18) hemidiaphragms from subjects who completed the entire intra-operative stimulation protocol. Insufficient tissue was available in two unstimulated hemidiaphragms. Tissue obtained from one participant contained large proportions of intramuscular fat that prevented a measurement.
Measure: Mean (Standard Deviation); unit: mU/mg protein
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 20 | 18
mU/mg protein | 0.175 (0.01) | 0.196 (0.01)

3. Primary Outcome: Lipid Peroxidation
Description: Lipid peroxidation will be assessed by measuring 4-hydroxy-2-nonenal-modified proteins. It will be quantified as arbitrary optical density units.
Time Frame: Up to eight hours
Population: Protein content was measured by traditional Western blot. Samples were analyzed from the stimulated and unstimulated hemidiaphragms of the first 11 participants. Protein quantification was normalized to total protein and optical density units of the stimulated and unstimulated hemidiaphragm were reported.
Measure: Mean (Standard Deviation); unit: Arbitrary optical density units (U)
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 11 | 11
Arbitrary optical density units (U) | 1.037 (0.145) | 1.061 (0.134)

4. Primary Outcome: Citrate Cynthase Activity
Description: Changes in electron transport chain will be assessed by measuring citrate cynthase activity. It will be quantified as nmol/mg protein/min.
Time Frame: Up to eight hours
Population: Citrate synthase activity was measured in the stimulated (n=20) and unstimulated (n=18) hemidiaphragms from subjects who completed the entire intra-operative stimulation protocol. Insufficient tissue was available in two unstimulated hemidiaphragms. Tissue obtained from one participant contained large proportions of intramuscular fat that prevented a measurement.
Measure: Mean (Standard Deviation); unit: nmol/mg protein/min
Arm/Group | Control | Stimulation
Number analyzed (Participants) | 18 | 20
nmol/mg protein/min | 0.084 (0.006) | 0.082 (0.004)

5. Primary Outcome: Single Diaphragm Fiber, Specific Force
Description: Specific force of single diaphragm fibers represents the force generated per unit area.
Time Frame: Up to eight hours
Population: Specific force represents force generation per cross sectional area of single diaphragm fibers and was calculated from an average of 10 slow and 10 fast single fibers obtained from each hemidiaphragm, per subject. Of the 21 patients who completed intraoperative stimulation procedures, single fiber measurements were not obtained in two participants due to unavailability of study personnel (n=2) and non-cardiac surgery (n=1).
Measure: Mean (Standard Error); unit: kN/m2
Units Other Than Participants: Muscle Fibers
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 18 | 18
Number analyzed (Muscle Fibers) | 372 | 373
kN/m2
  Slow Fibers: number analyzed (Muscle Fibers) | 186 | 196
  Slow Fibers | 102.64 (2.38) | 95.85 (4.62)
  Fast Fibers: number analyzed (Muscle Fibers) | 186 | 177
  Fast Fibers | 124.5 (2.39) | 126.93 (4.3)

6. Primary Outcome: Single Diaphragm Fiber, Rate of Tension Redevelopment
Description: Single diaphragm fiber mechanical force properties will be measured. The rate of tension redevelopment is quantified as s^(-1).
Time Frame: Up to eight hours
Population: Rate constant of tension development (ktr) represents the half-time of force recovery after release of a standardized stretch. ktr was calculated from an average of 10 slow and 10 fast single fibers obtained from each hemidiaphragm, per subject. Of the 21 patients who completed intraoperative stimulation procedures, single fiber measurements were not obtained in two participants due to unavailability of study personnel (n=2) and non-cardiac surgery (n=1).
Measure: Mean (Standard Error); unit: per second (force recovery rate)
Units Other Than Participants: Muscle Fibers
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 18 | 18
Number analyzed (Muscle Fibers) | 372 | 373
per second (force recovery rate)
  Slow Fibers: number analyzed (Muscle Fibers) | 186 | 196
  Slow Fibers | 1.102 (0.269) | 1.143 (0.236)
  Fast Fibers: number analyzed (Muscle Fibers) | 186 | 177
  Fast Fibers | 4.744 (1.322) | 4.777 (1.369)

7. Primary Outcome: Calcium Sensitivity (pCa50)
Description: The pCa50 value is the logarithmic scale of pCa (sensitivity of Ca+2) at which half-maximal force generation was obtained. The pCa value is calculated as the -log10[Ca (nm)]; the pCa50 is the -log10[Ca (nm)] at which half-maximal force is generated.
Time Frame: Up to eight hours
Population: pCa50 represents the sensitivity of pCa (concentration of Ca+2: -log10[Ca+2]) at which half-maximal force generation was obtained. It was calculated from an average of 10 slow and 10 fast single fibers obtained from each hemidiaphragm, per subject. Of the 21 patients who completed intraoperative stimulation procedures, single fiber measurements were not obtained in two participants due to unavailability of study personnel (n=2) and non-cardiac surgery (n=1).
Measure: Mean (Standard Error); unit: -log10[Ca2+]
Units Other Than Participants: Muscle Fibers
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 18 | 18
Number analyzed (Muscle Fibers) | 372 | 373
-log10[Ca2+]
  Slow Muscle Fibers: number analyzed (Muscle Fibers) | 186 | 196
  Slow Muscle Fibers | 5.805 (0.158) | 5.797 (0.161)
  Fast Muscle Fibers: number analyzed (Muscle Fibers) | 186 | 177
  Fast Muscle Fibers | 5.888 (0.115) | 5.887 (0.121)

8. Primary Outcome: Difference in Total Titin to Myosin Heavy Chain Ratio
Description: The quantities of total titin protein and myosin heavy chain protein content in homogenized diaphragm fiber specimens were measured and then calculated as a ratio of total titin to myosin heavy chain content (unitless value). The statistical approach was selected apriori as the difference of the ratio between the stimulated and unstimulated sides.
Time Frame: Up to eight hours
Population: The quantities of total titin protein and myosin heavy chain protein content in homogenized diaphragm fiber specimens were measured and then calculated as a ratio of total titin to myosin heavy chain content. The statistical approach selected to test the effect of stimulation on titin:myosin heavy chain ratio was selected apriori as the difference between the stimulated and unstimulated sides.
Measure: Mean (Standard Deviation); unit: Total titan/MHC Ratio
Groups:
- Control: No electrical stimulation of hemidiaphragm.
- Stimulated: Electrical stimulation of hemidiaphragm.
Arm/Group | Control | Stimulated
Number analyzed (Participants) | 11 | 11
Total titan/MHC Ratio | 0.111 (0.042) | 0.103 (0.044)

9. Primary Outcome: Difference in Titin Exon Composition
Description: The composition of titin exons will be assessed and quantified via real-time polymerase chain reaction (qPCR). The N2A and tT2 will be calculated as a percentage of total titin.
Time Frame: Up to eight hours
Population: The composition of the N2A and tT2 exons of the titin protein was obtained from homogenized tissue of the unstimulated and stimulated hemidiaphragms of the first 11 subjects. The relative abundance of each exon was calculated as a percentage of total titin.
Measure: Mean (Standard Deviation); unit: Percent of total titin
Arm/Group | Control | Stimulated
Number analyzed (Participants) | 11 | 11
Percent of total titin
  Percentage N2A | 96.1 (9.3) | 96.3 (6.9)
  Percentage tT2 | 3.9 (9.3) | 3.7 (6.9)

10. Primary Outcome: Difference in Titin Binding Protein Content
Description: The content of titin binding proteins will be quantified via Western blot. It will be normalized to a reference protein (GAPDH) and presented as optical intensity (AU).
Time Frame: Up to eight hours
Population: Content of titin binding proteins including MARP1 (ANKRD-1) and MARP2 (ANKRD-2) were measured in homogenized tissue obtained from the stimulated and unstimulated hemidiaphragms of the first 11 subjects and quantified using western blot. The results were normalized to the optical intensity of GAPDH (AU).
Measure: Mean (Standard Deviation); unit: AU
Groups:
- Stimulated: Electrical stimulated hemidiaphragms.
Arm/Group | Control | Stimulated
Number analyzed (Participants) | 11 | 11
AU
  ANKRD1 | 0.0165 (0.0279) | 0.0167 (0.025)
  ANKRD2 | 1.39 (0.44) | 1.28 (0.52)

11. Primary Outcome: Difference in Calpain 1 Protein Content
Description: Calpain 1 (mu-calpain) will be measured with Western Blot analysis and will be presented as percent of total intensity in stimulated and unstimulated hemidiaphragms
Time Frame: Up to eight hours
Population: Calpain-1 (µ-calpain) protein content was measured by traditional Western blot. Samples were analyzed from the stimulated and unstimulated hemidiaphragms of the first 9 participants and normalized to total protein. The statistical approach selected to test the effect of stimulation on oxidative stress-related protein content was selected apriori as the difference between the stimulated and unstimulated sides. Full-length (80kDa) and truncated (76 kDa) isoforms are reported.
Measure: Mean (Standard Deviation); unit: Percent of total Intensity
Arm/Group | Control | Stimulated
Number analyzed (Participants) | 11 | 11
Percent of total Intensity
  Full length (80 kDa) CLP1 isoform | 74 (5.4) | 72.4 (5.4)
  Truncated (76 kDa) CLP1 isoform | 14.1 (2.6) | 15 (3)

12. Primary Outcome: Difference in Calpain 2 Protein Content
Description: Calpain 2 will be measured with automated, capillary-based immunoassay using a Jess System, normalized to total protein, and will be presented as an area of corrected peak (AU) in stimulated and unstimulated hemidiaphragms.
Time Frame: Up to eight hours
Population: Protein content of AKT, p-AKT, calpain-2, calpain-3, caspase-3, atrogin-1 was measured by automated, capillary-based immunoassay using a Jess System. Samples were analyzed from the stimulated and unstimulated hemidiaphragms of the first 9 participants and normalized to total protein.
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Control | Stimulated
Number analyzed (Participants) | 11 | 11
AU | 274938 (118636) | 357182 (219400)

13. Primary Outcome: Difference in Calpain 3 Protein Content
Description: Calpain 3 will be measured with Western Blot analysis and will be presented as a ratio of cleaved to total calpain 3 (unitless value) in stimulated and unstimulated hemidiaphragms.
Time Frame: Up to eight hours
Population: Protein content of AKT, p-AKT, calpain-2, calpain-3, caspase-3, atrogin-1 was measured by automated, capillary-based immunoassay using a Jess System. Samples were analyzed from the stimulated and unstimulated hemidiaphragms of the first 9 participants and normalized to total protein. The statistical approach selected to test the effect of stimulation on oxidative stress-related protein was selected apriori as the difference between the stimulated and unstimulated sides.
Measure: Mean (Standard Deviation); unit: ratio of cleaved/total calpain 3
Arm/Group | Control | Stimulated
Number analyzed (Participants) | 11 | 11
ratio of cleaved/total calpain 3 | 2.98 (1.35) | 3.21 (1.9)

14. Primary Outcome: Difference in Caspase-3 Protein Content
Description: Caspase-3 will be measured with Western Blot analysis, normalized to total protein loaded in each lane, and will be presented as an area of corrected peak (AU) in stimulated and unstimulated hemidiaphragm muscle fibers.
Time Frame: Up to eight hours
Population: Protein content of calpain-2, calpain-3, caspase-3, atrogin-1 was measured by automated, capillary-based immunoassay using a Jess System. Samples were analyzed from the stimulated and unstimulated hemidiaphragms of the first 9 participants and normalized to total protein.
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Control | Stimulated
Number analyzed (Participants) | 11 | 11
AU | 274328 (70600) | 317726 (164524)

15. Primary Outcome: Atrogin 1
Description: Atrogin 1 will be measured with Jess protein immunoassay analysis, normalized to total protein, and will be presented as the corrected peak area (AU) in stimulated and unstimulated hemidiaphragm muscle fibers.
Time Frame: Up to eight hours
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: AU
Groups:
- Stimulated: No electrical stimulation of hemidiaphragm.
Arm/Group | Control | Stimulated
Number analyzed (Participants) | 11 | 11
AU | 634046 (377885) | 675965 (379914)

16. Other Pre Specified Outcome: Mitochondrial Reactive Oxygen Species Production
Description: Mitochondrial reactive oxygen species (ROS) production will be assessed using an in situ approach to measure hydrogen peroxide production in permeabilized diaphragm skeletal muscle fiber bundles. It will be quantified as pmol/min/mg dry weight.
Time Frame: Up to eight hours
Population: Limited tissue quantity did not permit analysis.
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Cytochrome c Oxidase (COX) Activity
Description: Changes in electron transport chain will be assessed by measuring cytochrome c oxidase (COX) activity. It will be quantifed as Units/mcg protein.
Time Frame: Up to eight hours
Population: Limited tissue quantity did not permit analysis.
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 0 | 0

18. Other Pre Specified Outcome: Nuclear DNA Mutation Frequency
Description: Long-Amplicon quantitative PCR will be used to measure the frequency of nuclear DNA mutations. It will be quantified as number of lesions/10 kilobases.
Time Frame: Up to eight hours
Population: Limited tissue quantity did not permit analysis.
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 0 | 0

19. Other Pre Specified Outcome: Titin Size
Description: Titin integrity will be assessed. A relative titin size will be quantified in nm.
Time Frame: Up to eight hours
Population: Limited tissue quantity did not permit analysis.
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 0 | 0

20. Other Pre Specified Outcome: Caspase-9
Description: Caspase-9 will be measured with Western Blot anaylsis and will be presented as percent difference in expression.
Time Frame: Up to eight hours
Population: Changes in Caspase-9 protein were not evaluated due to lack of a reliable antibody with preparatory validation studies.
Groups:
- Difference Between Groups: The percentage difference in protein, between the stimulated and unstimulated/control hemidiaphragms.
Arm/Group | Difference Between Groups
Number analyzed (Participants) | 0

21. Other Pre Specified Outcome: 20S Proteasome
Description: 20S proteasome will be measured with Western Blot anaylsis and will be presented as percent difference in expression.
Time Frame: Up to eight hours
Population: Changes in 20S proteasome protein were not evaluated due to lack of a reliable antibody with preparatory validation studies.
Arm/Group | Difference Between Groups
Number analyzed (Participants) | 0

22. Other Pre Specified Outcome: 26S Proteasome
Description: 26S proteasome will be measured with Western Blot anaylsis and will be presented as percent difference in expression.
Time Frame: Up to eight hours
Population: Changes in 26S Proteasome protein were not evaluated due to lack of a reliable antibody with preparatory validation studies.
Arm/Group | Difference Between Groups
Number analyzed (Participants) | 0

23. Other Pre Specified Outcome: 28SrRNA
Description: 28SrRNA will be measured with Western Blot anaylsis and will be presented as percent difference in expression.
Time Frame: Up to eight hours
Population: Differences in 28SrRNA were not completed due to challenges with cross-species validation of reagents and reference values.
Arm/Group | Difference Between Groups
Number analyzed (Participants) | 0

24. Other Pre Specified Outcome: 18SrRNA
Description: 18SrRNA will be measured with Western Blot anaylsis and will be presented as percent difference in expression.
Time Frame: Up to eight hours
Population: Differences in 18SrRNA were not completed due to challenges with cross-species validation of reagents and reference values.
Arm/Group | Difference Between Groups
Number analyzed (Participants) | 0

25. Other Pre Specified Outcome: Foxo-3
Description: Foxo-3 will be measured with Western Blot anaylsis and will be presented as percent difference in expression.
Time Frame: Up to eight hours
Population: Changes in Foxo-3 protein were not evaluated due to lack of a reliable antibody with preparatory validation studies.
Arm/Group | Difference Between Groups
Number analyzed (Participants) | 0

26. Other Pre Specified Outcome: 45S Pre-rRNA
Description: 45S pre-rRNA will be measured with Western Blot anaylsis and will be presented as percent difference in expression.
Time Frame: Up to eight hours
Population: Changes in 45S pre-rRNA protein were not evaluated due to lack of a reliable antibody with preparatory validation studies.
Arm/Group | Difference Between Groups
Number analyzed (Participants) | 0

27. Other Pre Specified Outcome: Mitochondrial DNA Mutation Frequency
Description: Long-Amplicon quantitative PCR will be used to measure the frequency of mitochondrial DNA mutations. It will be quantified as number of lesions/10 kilobases.
Time Frame: Up to eight hours
Population: Limited tissue quantity did not permit analysis.
Arm/Group | Stimulation | Control
Number analyzed (Participants) | 0 | 0

28. Other Pre Specified Outcome: MurF1
Description: MurF1 will be measured with Western Blot anaylsis and will be presented as percent difference in expression.
Time Frame: Up to eight hours
Population: Changes in MuRF1 protein were not evaluated due to lack of a reliable antibody with preparatory validation studies.
Arm/Group | Difference Between Groups
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From enrollment of each patient until their hospital discharge, which was typically within 7-10 days post-op.
Description: Standard CT.gov definitions were used, and assessments were conducted systematically through the medical record and consultation with the study surgeons.
Arm/Group | Participants Undergoing Elective, Open Cardiothoracic Surgical Procedures Lasting 4 Hours or Greater
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 14/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Undergoing Elective, Open Cardiothoracic Surgical Procedures Lasting 4 Hours or Greater (N=21)
Arrhythmias (Cardiac disorders) | 10 (11)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Dysphagia (General disorders) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Methycillin sensitive staph aureus infection (Infections and infestations) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Near-syncope (Cardiac disorders) | 1 (1)
Low cardiac index (Cardiac disorders) | 1 (1)
Sternal wound infection (Infections and infestations) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Acute MCA stroke (Vascular disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Sternal malunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Undergoing Elective, Open Cardiothoracic Surgical Procedures Lasting 4 Hours or Greater (N=21)
Postoperative Pain (General disorders) | 20 (20)
Anemia (Blood and lymphatic system disorders) | 17 (17)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (10)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Leukocytosis (Blood and lymphatic system disorders) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Hypotension (Vascular disorders) | 4 (4)
Bradycardia (Cardiac disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bilateral lower extremity edema (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03303040/Prot_SAP_000.pdf